CLINICAL TRIAL: NCT00824252
Title: Spousal Support, Emotional Disclosure, and Adjustment to Head and Neck Cancer
Brief Title: Spousal Support in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008-0188; K07CA124668 (NIH)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Head And Neck Cancer
Keywords: Head And Neck Cancer; HNC; Radiation Therapy; Spousal Support; Emotional Disclosure; Observational; Social Constraints; Questionnaires; Videotaped Interview; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spousal Support: Questionnaire for Head and Neck Cancer Patients + Spouses
  Interventions: Behavioral: Questionnaires & Study Visit

INTERVENTIONS:
Behavioral: Questionnaires & Study Visit — Individual Questionnaires (1 hour) and videotaped discussion during Study Visit (1 1/4 hours)
  Other Names: Survey

SUMMARY:
The goal of this research study is to look at social and relationship factors that may affect the quality of life of patients with head and neck cancer and their spouses.

DETAILED DESCRIPTION:
If you agree to take part in this study, you first fill out a questionnaire, which will take about 1 hour. You will also have a study visit with your spouse, where you and your spouse will fill out several questionnaires, have a videotaped discussion, and complete tasks on the computer. This study visit will last about 75 minutes.

Health and Relationship Questionnaire:

On Day 1 you will be given a questionnaire about your health and your relationship with your spouse. This will be before you begin treatment. You may complete the questionnaire while waiting for your clinic appointment, or you may take it home, complete it, and return it by mail. It will take about 60 minutes to complete.

If you agree to take part in this study, your spouse will also be asked to take part. If your spouse does not wish to take part, your participation in this study will be over after you complete the questionnaire.

Study Visit:

During the first 2 weeks after you start treatment, you and your spouse will come to the clinic together for a study visit. The visit will take about 75 minutes. For all of the procedures at this visit, you and your spouse will be in the same room together. A study staff member will also be in the room, except for during the videotaped discussions. The following procedures will be performed at the study visit:

* You will complete a questionnaire that asks you to identify one instance where you felt supported by your spouse since the cancer diagnosis, and one issue that has caused conflict with your spouse since the cancer diagnosis. You will also complete a questionnaire about your mood. Your spouse will complete the same questionnaires. This will take about 10-15 minutes.
* You and your spouse will take part in a videotaped discussion. You will discuss the topic you identified as an instance where you felt supported by your spouse since the cancer diagnosis. Your spouse will also discuss the topic he/she identified as an instance where he/she felt supported by you since the cancer diagnosis. This will take about 10-15 minutes.
* After the discussion, you and your spouse will be asked to complete a cognitive (thinking) task, on separate computers. Words in different colors will appear on the computer screen. The goal of the task is to name the color of the words, as quickly as possible. It will take about 5 minutes to complete the task.
* After the cognitive task, you and your spouse will complete separate questionnaires that will ask questions about the discussion and how you feel about it. This will take about 5-10 minutes.
* You and your spouse will take part in another videotaped discussion. This time, you will discuss the topic you identified as causing conflict with your spouse since the cancer diagnosis. Your spouse will also discuss the topic he/she identified as causing conflict since the cancer diagnosis. It will take about 10-15 minutes.
* After the discussion, you and your spouse will repeat the same cognitive task. It will again be on separate computers and will take about 5 minutes.
* After the cognitive task, you and your spouse will complete separate questionnaires that will ask questions about the discussion and how you feel about it. This will take about 5-10 minutes.
* At the conclusion of the study visit, you will have the option to view the videotape of your discussion with your spouse. If, after viewing your videotape you decide for any reason that you do not want it to be used for research, the tape will be destroyed.

Follow-Up Questionnaire:

You will complete the Health and Relationship questionnaire 2 more times.

If possible, you will complete this questionnaire while you are at the clinic for your regularly scheduled follow-up visits that will occur 4 months and 12 months after you complete your radiation treatment. Otherwise, if your appointment is not on the same schedule as this study's questionnaire schedule, you will receive the questionnaire by mail and you should mail it back to the study staff.

Information Collection:

During the course of this study, a study staff member will review your medical records to collect medical information such as your diagnosis and health history.

Length of Study:

After you complete the last questionnaire (Month 12), your participation in this study will be over.

This is an investigational study. For any questionnaires that you are asked to return by mail, you will be provided stamped envelopes.

Up to 452 participants (226 patients and 226 spouses) will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Part 2. Patient is initiating radiation therapy for newly diagnosed head and neck cancer
2. Part 2. Patient has an Eastern Cooperative Oncology Group performance status score of 2 or less
3. Part 2. Patient has a spouse or significant other with whom he/she resides
4. Part 2. Patient is able to vocalize well enough to complete the spousal interaction task
5. Parts 1 and 2. Patient and spouse are able to read and speak English
6. Parts 1 and 2. Patient and spouse are able to provide informed consent
7. Parts 1 and 2. Patient and spouse are at least 18 years of age
8. Part 1. Individual is a patient who was diagnosed with head and neck cancer or the spouse or partner of an patient who was diagnosed with head and neck cancer and resides with the patient.

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer patients who will be starting radiation therapy and their spouses.
Sampling Method: Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2008-12-08 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Social + Relationship Factors Affecting QOL of HNC Patients & Spouses | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, PHD, MA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org